CLINICAL TRIAL: NCT00942994
Title: An 8-week Multicenter, Randomized, Double-blind, Active Controlled, Parallel Group, Forced Titration Study to Evaluate the Efficacy and Safety of Aliskiren/Amlodipine/HCTZ Compared to Aliskiren/Amlodipine in US Minority Patients With Stage 2 Hypertension
Brief Title: Aliskiren/Amlodipine/Hydrochlorothiazide (HCTZ) Versus Aliskiren/Amlodipine in US Minority Patients With Stage II Systolic Hypertension
Acronym: ASCENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPA100AUS02
Record Dates: First submitted 2009-07-19; First posted 2009-07-21 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Hypertension; Aliskiren; Amlodipine; HCTZ; Systolic blood pressure; Diastolic blood pressure; Stage II; Combination
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Triple Therapy (Aliskiren/Amlodipine/HCTZ) (Experimental): At week 0 patients were randomized to aliskiren/amlodipine 150/5 mg. At week 1, patients were force titrated to aliskiren/amlodipine/HCTZ 150/5/12.5 mg. At week 2, patients were force titrated to aliskiren/amlodipine/HCTZ 300/5/25 mg. At week 4, patients were force titrated to aliskiren/amlodipine/HCTZ 300/10/25 mg.
  Interventions: Drug: Aliskiren/Amlodipine and Hydrochlorothiazide (HCTZ)
- Dual Therapy (Aliskiren/Amlodipine) (Active Comparator): At week 0 patients were randomized to amlodipine 5 mg. At week 1, patients were force titrated to aliskiren/amlodipine 150/5 mg. At week 2, patients were force titrated to aliskiren/amlodipine 300/5 mg. At week 4, patients were force titrated to aliskiren/amlodipine 300/10 mg.
  Interventions: Drug: Aliskiren/Amlodipine

INTERVENTIONS:
Drug: Aliskiren/Amlodipine — Amlodipine capsule (5 mg)
  Aliskiren/Amlodipine tablets (150/5 mg, 300/5 mg, 300/10 mg)
  Arms: Dual Therapy (Aliskiren/Amlodipine)
Drug: Aliskiren/Amlodipine and Hydrochlorothiazide (HCTZ) — Aliskiren/Amlodipine tablets (150/5 mg, 300/5 mg, 300/10 mg)
  HCTZ capsule (12.5 mg, 25mg)
  Arms: Triple Therapy (Aliskiren/Amlodipine/HCTZ)

SUMMARY:
The purpose of the study is to compare the combination of aliskiren, amlodipine and Hydrochlorothiazide (HCTZ) versus the combination of aliskiren and amlodipine as therapy in minority Stage 2 hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly diagnosed or have a history of hypertension, who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Men or women 18 years and older of minority background; self-identified.
* Patients with stage 2 hypertension defined as MSSBP ≥160 mmHg and <200 mmHg at Visit 5 (randomization).

Exclusion Criteria:

* Patients with MSDBP ≥110 mmHg and/or MSSBP ≥200 mmHg as measured by office cuff at any visit.
* Patients on 4 or more antihypertensive medications.
* Patients with uncontrolled hypertension (MSSBP >180 mmHg) taking more than 1 antihypertensive medication at Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (5):
- United States (5):
  - K and S Research Services, Little Rock, Arkansas
  - Well Pharma Medical Research, South Miami, Florida
  - Hyde Park Health Associates, Mattapan, Massachusetts
  - Manassas Clinical Research Center, Manassas, Virginia
  - Scriber Kidney Center, Seattle, Washington

REFERENCES:
- [Result] Ferdinand KC, Weitzman R, Israel M, Lee J, Purkayastha D, Jaimes EA. Efficacy and safety of aliskiren-based dual and triple combination therapies in US minority patients with stage 2 hypertension. J Am Soc Hypertens. 2011 Mar-Apr;5(2):102-13. doi: 10.1016/j.jash.2011.01.006. PMID 21414565
- [Derived] Ferdinand KC, Weitzman R, Purkayastha D, Sridharan K, Jaimes EA. Aliskiren-based dual- and triple-combination therapies in high-risk US minority patients with stage 2 hypertension. J Am Soc Hypertens. 2012 May-Jun;6(3):219-27. doi: 10.1016/j.jash.2011.12.002. Epub 2012 Feb 3. PMID 22305998

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren / Amlodipine / HCTZ: At week 0 patients were randomized to aliskiren/amlodipine 150/5 mg. At week 1, patients were force titrated to aliskiren/amlodipine/HCTZ 150/5/12.5 mg. At week 2, patients were force titrated to aliskiren/amlodipine/HCTZ 300/5/25 mg. At week 4, patients were force titrated to aliskiren/amlodipine/HCTZ 300/10/25 mg.
- Aliskiren / Amlodipine: At week 0 patients were randomized to amlodipine 5 mg. At week 1, patients were force titrated to aliskiren/amlodipine 150/5 mg. At week 2, patients were force titrated to aliskiren/amlodipine 300/5 mg. At week 4, patients were force titrated to aliskiren/amlodipine 300/10 mg.
Period: Overall Study
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Started | 203 | 209
Completed | 187 | 190
Not Completed | 16 | 19
Not completed — Adverse Event | 7 | 4
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 1
Not completed — Patient withdrew consent | 5 | 8
Not completed — Lost to Follow-up | 1 | 4
Not completed — Protocol deviation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine | Total
Number analyzed (Participants) | 202 | 209 | 411
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline characteristics are given for Safety Set. The Safety Set included all patients who received at least one dose of double-blind trial medication. One patient was excluded from the Safety Set because the patient was withdrawn from the study without receiving any dose of study medication.
  years | 55.7 (9.79) | 54.7 (10.19) | 55.2 (10.00)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are given for Safety Set. The Safety Set included all patients who received at least one dose of double-blind trial medication. One patient was excluded from the Safety Set because the patient was withdrawn from the study without receiving any dose of study medication.
  Participants
    Female | 107 | 100 | 207
    Male | 95 | 109 | 204

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 8
Description: To evaluate change from baseline in MSSBP after 8 weeks of treatment with an aliskiren, amlodipine, and HCTZ treatment regimen versus an aliskiren and amlodipine treatment regimen in minority patients with Stage 2 hypertension.
Time Frame: Baseline and week 8
Population: Analysis was based on the Full Analysis Set consisting of all patients to whom study medication had been assigned. Last-observation-carried-forward was used. Baseline was not carried forward. In the Aliskiren/Amlodipine/HCTZ group, 5 patients did not have a post baseline measure. Hence, change from baseline to week 8 is reported for 197 patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
mmHg
  Baseline [N=202, 209] | 167.08 (7.277) | 167.41 (7.118)
  Week 8 [N=197, 209] | 130.73 (13.06) | 137.87 (16.013)
  Change from baseline to week 8 [N=197, 209] | -36.43 (13.904) | -29.54 (15.674)

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 8
Description: To evaluate change from baseline in MSDBP after 8 weeks of treatment with an aliskiren, amlodipine, and HCTZ treatment regimen versus an aliskiren and amlodipine treatment regimen in minority patients with Stage 2 hypertension.
Time Frame: Baseline and week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
mmHg
  Baseline [N=202, 209] | 95.25 (8.985) | 95.25 (8.342)
  Week 8 [N=197, 209] | 80.10 (10.317) | 83.17 (10.116)
  Change from baseline to week 8 [N=197, 209] | -15.10 (9.707) | -12.08 (9.062)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control (Defined as MSSBP < 140 mmHg and MSDBP < 90 mmHg) During 8 Weeks
Description: To evaluate the cumulative percentage of patients achieving Blood Pressure control (defined as patients achieving an MSSBP <140 mmHg and MSDBP <90 mmHg) during 8 weeks of treatment with an aliskiren, amlodipine, and HCTZ treatment regimen versus an aliskiren and amlodipine treatment regimen in minority patients with Stage 2 hypertension. Cumulative refers to achieving BP control before or at the corresponding visit.
Time Frame: 8 weeks
Population: Analysis was based on the Full Analysis Set (FAS) consisting of all patients to whom study medication had been assigned.
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
Percentage of Participants
  Week 2 | 50.5 | 40.2
  Week 4 | 74.8 | 57.4
  Week 8 | 81.7 | 67.9

4. Secondary Outcome: Percentage of Responders (Defined as Patients With MSSBP < 140 mmHg or a Reduction From Baseline in MSSBP of ≥20 mmHg) During 8 Weeks.
Description: To compare the cumulative percentage of responders (defined as patients with MSSBP <140 mmHg or a decrease from baseline ≥20 mmHg) during 8 weeks of treatment with an aliskiren, amlodipine, and HCTZ treatment regimen versus an aliskiren and amlodipine treatment regimen in minority patients with Stage 2 hypertension. Cumulative refers to achieving a response before or at the corresponding visit.
Time Frame: 8 weeks
Population: Analysis was based on the Full Analysis Set (FAS) consisting of all patients to whom study medication had been assigned.
Measure: Number; unit: Percentage of Responders
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
Percentage of Responders
  Week 2 | 79.2 | 72.2
  Week 4 | 91.1 | 84.7
  Week 8 | 92.6 | 91.9

5. Other Pre Specified Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP) at Week 2 and Week 4
Description: Primary objective at additional timepoint.
Time Frame: Baseline, Week 2 and Week 4
Population: Analysis was based on the Full Analysis Set consisting of all patients to whom study medication had been assigned. Last-observation-carried-forward was used. Baseline was not carried forward. In the Aliskiren/Amlodipine/HCTZ group, 5 patients did not have a post baseline measure. Hence, change from baseline is reported for 197 patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
mmHg
  Baseline [N=202, 209] | 167.08 (7.277) | 167.41 (7.118)
  Week 2 [N=197, 209] | 138.35 (12.578) | 143.77 (13.922)
  Change from baseline to week 2 [N=197, 209] | -28.81 (12.640) | -23.64 (13.673)
  Week 4 [N=197, 209] | 132.42 (12.027) | 140.43 (13.961)
  Change from baseline to week 4 [N=197, 209] | -34.74 (12.145) | -26.98 (13.389)

6. Other Pre Specified Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP) at Week 2 and Week 4
Description: Secondary objective at additional timepoint.
Time Frame: Baseline, Week 2 and Week 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Number analyzed (Participants) | 202 | 209
mmHg
  Baseline [N=202, 209] | 95.25 (8.985) | 95.25 (8.342)
  Week 2 [N=197, 209] | 84.26 (9.597) | 86.24 (8.908)
  Change from baseline to week 2 [N=197, 209] | -10.95 (8.569) | -9.01 (7.872)
  Week 4 [N=197, 209] | 81.29 (9.177) | 85.35 (9.567)
  Change from baseline to week 4 [N=197, 209] | -13.92 (8.891) | -9.91 (7.606)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: AEs were analyzed in the Safety Set. The Safety Set included all patients who received at least one dose of double-blind trial medication. One patient was excluded from the Safety Set because the patient was withdrawn from the study without receiving any dose of study medication.
Arm/Group | Aliskiren / Amlodipine / HCTZ | Aliskiren / Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/202 | 3/209
Other Adverse Events (participants affected / at risk) | 22/202 | 18/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Amlodipine / HCTZ (N=202) | Aliskiren / Amlodipine (N=209)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren / Amlodipine / HCTZ (N=202) | Aliskiren / Amlodipine (N=209)
Headache (Nervous system disorders) | 22 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.